CLINICAL TRIAL: NCT06737432
Title: Respiratory Knowledge Portal Application to Reduce Ventilator Associated Events, Ventilator Induced Lung Injury and Alarm Parameter Variance
Brief Title: Respiratory Knowledge Portal Computer and Phone Application to Improve Quality of Mechanical Ventilation by Reducing the Number of Ventilator Associated Events, Injury Created by the Ventilator and Unsafe Setting of Alarms.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Vyaire Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0313
Record Dates: First submitted 2024-07-11; First posted 2024-12-17 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Ventilation; ARDS; Respiratory Failure; Mechanical Ventilation; Ventilator-induced Lung Injury (VILI); Quality Improvement; Ventilator Associated Events
Keywords: Computer aided mechanical ventilation; Mechanical ventilation quality; Mechanical ventilation; Mechanical ventilation safety; Ventilator monitoring application
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency; Ventilator-Induced Lung Injury

STUDY DESIGN:
Masking Description: Monitoring 3-4 months prior to intervention or use of the software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): We will monitor without clinician use of the software.
- Use of RKP (Active Comparator): Use of RKP alerts to the standard of care.
  Interventions: Other: RKP Monitoring Software

INTERVENTIONS:
Other: RKP Monitoring Software — Use of RKP alerting and monitoring software.
  Arms: Use of RKP

SUMMARY:
Ventilator associated events (VAE) is a quality metric defined by 48 hours of stability followed by 48 hours of escalation of ventilator settings within the ICU. VAE have been associated with poor outcomes and increases the cost of care, yet is not easy to avoid. Operationalizing all the standards of care known to improve outcomes of those requiring mechanical ventilation in the critical care environment requires a comprehensive approach. ICU teams are encouraged to follow best practice protocols to help liberate and prevent VAEs. Yet, compliance with protocols in most ICUs is suboptimal for multiple reasons. With the advent of computerized mechanical ventilators capable of streaming data from breath to breath and biomedical integration systems (BMDI) such as Capsule (UTMB's BMDI system), software systems have been developed to help identify variances in the standard of care. Automation in near real-time ventilator data feedback has been shown to reduce the incidences of VAEs.

This quality improvement project will leverage Vyaire's Respiratory Knowledge Portal (RKP) to collect and store meaningful data regarding ventilator-associated events (VAE), alarm policy compliance, ventilator weaning, and lung protective analytics.

Goals:

1. To collect quality metrics utilizing RKP from patients requiring mechanical ventilation over a 3-4-month period for a retrospective baseline analysis.
2. Provide the RKP tool to the ICU team to determine if the use of RKP's webportal and Messenger Zebra phone app improves quality of mechanical ventilation and outcomes.
3. To determine a return on investment (ROI) for a software system like RKP.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects requiring invasive mechanical ventilation.
2. Subjects is in one of the monitored Galveston campus ICUs.
3. Ages 0-100

Exclusion Criteria:

1. Is in an ICU not monitored by RKP.
2. Adults on high frequency ventilation (pediatric patients are NOT excluded).
3. Any patient requiring ECMO.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Ventilator-Associated Events | 3-4 months

SECONDARY OUTCOMES:
Number of Ventilator Alarm Set Outside of Compliance | 3-4 months
  Ventilator alarms set by the RT
Duration of Days on mechanical ventilation | 3-4 months
  Does the weaning of mechanical ventilation improve through the measurements of spontaneous breathing trials.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No